CLINICAL TRIAL: NCT02684786
Title: A Phase I Study of Stellate Ganglion Block and / or Reserpine in Group 2 Pulmonary Hypertension
Brief Title: A Study of Stellate Ganglion Block and / or Reserpine in Group 2 Pulmonary Hypertension
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: IRB did not approve
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Joseph L. Blackshear, Consultant, Department of Cardiovascular Diseases, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-000928
Record Dates: First submitted 2016-02-04; First posted 2016-02-18 (Estimated); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Pulmonary Artery Hypertension
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension | interventions — Reserpine; Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prior right heart catheterization (Experimental): Patients with qualifying hemodynamics from prior right heart catheterization will receive open label reserpine, 0.05 mg by mouth daily for two weeks, then 0.10 mg by mouth daily for two weeks, and then have repeat non-invasive assessments of status.
  Interventions: Drug: reserpine
- Scheduled for right heart catheterization (Experimental): Patients with suspected group 2 pulmonary hypertension by clinical and non-invasive assessments and are scheduled to undergo clinically indicated right heart catheterization will have pulmonary artery pressures measured. If qualifying severity of group 2 pulmonary hypertension is present, after clinically indicated assessment of inhaled nitric oxide, their baseline hemodynamics will be allowed to re-equilibrate over 10 minutes, and then ultrasound guided left stellate ganglion block with lidocaine will be performed, and hemodynamics reassessed 10 minutes afterward
  Interventions: Procedure: stellate ganglion block; Drug: lidocaine

INTERVENTIONS:
Drug: reserpine — Patients with qualifying hemodynamics from prior right heart catheterization will receive open label reserpine, 0.05 mg by mouth daily for two weeks, then 0.10 mg by mouth daily for two weeks, and then have repeat non-invasive assessments of status
  Arms: Prior right heart catheterization
Procedure: stellate ganglion block — Patients with suspected group 2 pulmonary hypertension by clinical and non-invasive assessments and are scheduled to undergo clinically indicated right heart catheterization will have pulmonary artery pressures measured. If qualifying severity of group 2 pulmonary hypertension is present, after clinically indicated assessment of inhaled nitric oxide, their baseline hemodynamics will be allowed to re-equilibrate over 10 minutes, and then ultrasound guided left stellate ganglion block with lidocaine will be performed, and hemodynamics reassessed 10 minutes afterward
  Arms: Scheduled for right heart catheterization
Drug: lidocaine — Patients with suspected group 2 pulmonary hypertension by clinical and non-invasive assessments and are scheduled to undergo clinically indicated right heart catheterization will have pulmonary artery pressures measured. If qualifying severity of group 2 pulmonary hypertension is present, after clinically indicated assessment of inhaled nitric oxide, their baseline hemodynamics will be allowed to re-equilibrate over 10 minutes, and then ultrasound guided left stellate ganglion block with lidocaine will be performed, and hemodynamics reassessed 10 minutes afterward
  Arms: Scheduled for right heart catheterization

SUMMARY:
Pulmonary hypertension Group 2 (PH 2) associated with left-sided heart disease is relatively common, is associated with a poor prognosis, and unfortunately there are no proven medical treatments beyond attempts at correcting the left sided heart disease. Many PH 2 patients have evidence of active constriction of blood vessels from increased nerve traffic. Use of agents or procedures which produce a reversible chemical blockage of this nerve traffic have not been systematically tested in PH 2. The investigators will test whether acute interruption of sympathetic nervous system tone, which local anesthetic block of the stellate ganglion in the neck, will improve PH2, and also test whether the high blood pressure drug reserpine, which blocks sympathetic nerve activity, will do so during a one month trial period.

DETAILED DESCRIPTION:
Background. Pulmonary hypertension Group 2 (PH 2) associated with left-sided heart disease is relatively common, is associated with a poor prognosis, and unfortunately there are no proven medical treatments beyond attempts at correcting the left sided heart disease. Many PH 2 patients have evidence of vasoconstriction and increased sympathetic nervous system activity. Use of agents or procedures which produce a reversible chemical sympathectomy have not been systematically tested in PH 2.

Methods. Two groups will be eligible for participation: Group 1 (n=10): Patients with PH 2 previously documented by echocardiography (echo), 6 minute walk test, biomarkers, and right heart catheterization (RHC) will receive reserpine, 0.05 mg per day for two weeks, then, 0.1 mg per day for an additional two weeks. After one month, patients will be reassessed for New York Heart Association (NYHA) class and drug side effects, echocardiography, 6 minute walk assessment, and brain natriuretic peptide (BNP). Group 2 patients (n=10) will have clinically suspected PH 2 and be scheduled to undergo clinically indicated RHC. If during RHC PH 2 is confirmed, after assessment of nitric oxide responsiveness, their baseline hemodynamics will be re-established over 10 minutes, and a left stellate ganglion block with lidocaine will be performed, and immediate hemodynamic responsiveness assessed. Four hours post-procedure, a side effect questionnaire will be obtained. Group 2 patients who complete RHC will then begin reserpine treatment in the same manner as Group I patients.

Hypothesis and Impact. PH 2 is the most common type of pulmonary hypertension. The current diagnostic and therapeutic strategy aims to treat the left sided heart disease in attempt to normalize pulmonary artery pressure. The place of selective pulmonary vasodilators is undefined. The investigator's approach addresses inhibition of adverse pulmonary vasoconstriction mediated by the sympathetic nervous system in PH 2.

ELIGIBILITY:
Inclusion criteria:

* Prior right heart catheterization, with mean pulmonary artery pressure > 25 mm Hg, pulmonary capillary wedge pressure > 15 mm Hg, and diastolic pressure gradient (pulmonary artery diastolic pressure - mean pulmonary capillary wedge pressure) ≥ 7 mm Hg OR clinically suspected group 2 pulmonary hypertension from non-invasive testing with planned right heart catheterization (RHC).
* On stable diuretic therapy
* Able to attend end-study visit 4 weeks after study entry

Exclusion criteria:

* Anticipated surgery to correct heart lesion responsible for pulmonary hypertension
* Need for heparinization for right heart catheterization (not standard practice, but sometimes utilized)
* History of depression, or treatment with tricyclic anti-depressant, serotonin uptake inhibitor, monamine oxidase inhibitor
* Severe renal or hepatic impairment, creatinine clearance < 30 ml/minute or renal replacement therapy or post-kidney transplant, abnormal liver function with elevated enzymes> 1.5 times the upper limit of normal or prior liver transplant.
* Systolic blood pressure <100 mm Hg
* Heart rate < 60 beats per minute
* Inability to independently complete telephone follow-up at two weeks, and clinic end-study visit at 4 weeks.
* Pulmonary edema
* Infiltrative cardiomyopathy - amyloidosis
* Symptomatic orthostatic hypotension
* Women of childbearing age who have not had surgical sterilization and are not using oral contraceptives, or who's spouse has not had surgical sterilization will be excluded due to the length of the trial and the possibility that they could become pregnant after entry.
* Uncontrolled heartburn
* Prior surgery to the left neck, for example, carotid endarterectomy, or other surgery which would increase the risk of stellate ganglion block
* Known sensitivity, allergy, or contraindication to lidocaine, any local anesthetic, or reserpine

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | one month
  Adverse events of interest are for stellate ganglion block: pulmonary edema, bradycardia requiring treatment, hypotension requiring treatment, arrhythmia, pneumothorax, hoarseness, dysphagia, globus, left upper extremity weakness. For reserpine, heart failure hospitalization, syncope, all cause hospitalization, bradycardia requiring treatment, hypotension requiring treatment, new arrhythmia, edema requiring an increase in diuretics, depression, lethargy, nasal stuffiness, dizziness, orthostatic hypotension, falls, nightmares, sexual dysfunction, anxiety, dyspepsia.
  Adverse events classed as serious:
  * Life threatening serious adverse events including acute coronary syndrome with active ischemia, fatal arrhythmias, myocardial infarction, acute kidney injury, cardiogenic shock, stroke, pulmonary embolization, arterial and/or venous thrombosis, systemic embolization, severe hypotension, respiratory failure and death
  * Prolonged hospitalization or rehospitalization

SECONDARY OUTCOMES:
Number of participants with successful stellate ganglion block | One hour
  Stellate block: frequency of the occurrence of ptosis and conjunctival flushing.
Effect of stellate ganglion block on heart rate | One hour
  Heart rate before and after stellate ganglion block
Change in 6 minute walk distance from one month of reserpine therapy | One month
  Six minute walk distance, meters, baseline compared to one month
Change in brain natriuretic peptide (BNP) from one month of reserpine therapy | One month
  BNP, pg/ml, baseline compared to one month
Change in Doppler derived mean pulmonary artery pressure from one month of reserpine therapy | One month
  Mean pulmonary artery pressure estimate, mm Hg
Change in blood pressure from one month of reserpine therapy | One month
  Blood pressure, mm Hg, baseline versus one month
Change in Minnesota Living with heart failure questionnaire from one month of reserpine therapy | One month
  Minnesota Living with heart failure questionnaire aggregate score, baseline versus one month
Hemodynamic effect of stellate ganglion block | One hour
  Blood pressure, mm Hg, before and after stellate ganglion block
Hemodynamic effect of stellate ganglion block | One hour
  Pulmonary artery pressure, mm Hg, before and after stellate ganglion block
Hemodynamic effect of stellate ganglion block | One hour
  Pulmonary capillary wedge pressure, mm Hg, before and after stellate ganglion block
Hemodynamic effect of stellate ganglion block | One hour
  right atrial pressure, mm Hg, before and after stellate ganglion block
Hemodynamic effect of stellate ganglion block | One hour
  Cardiac output, liters per minute, before and after stellate ganglion block
Change in heart rate from one month of reserpine therapy | One month
  Heart rate, baseline versus one month

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Blackshear, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials